CLINICAL TRIAL: NCT01039961
Title: Evaluation of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Intravenous Dose(s) and a Single Oral Dose of GW856553 in Healthy Volunteers
Brief Title: PK Study of IV Formulation of GW856553
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113022
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Disease
Keywords: healthy volunteers; IV formulation study
MeSH Terms: conditions — Cardiovascular Diseases | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 mg IV (Experimental): Unit Dose Strength: 0.4 mg/mL
  Interventions: Drug: losmapimod 1 mg
- ?mg IV (Experimental): dose to be determined based on PK of first IV dose
  Interventions: Drug: losmapimod
- 15 mg (oral) (Experimental): two 7.5 mg tablets
  Interventions: Drug: losmapimod 15 mg

INTERVENTIONS:
Drug: losmapimod 1 mg — IV infusion
  Arms: 1 mg IV
Drug: losmapimod — IV infusion (dose to be determined based on PK from first dose)
  Arms: ?mg IV
Drug: losmapimod 15 mg — oral, two 7.5 mg tablets
  Arms: 15 mg (oral)

SUMMARY:
The purpose of this study is to evaluate the safety of an IV infusion of GW856553 in healthy volunteers.

DETAILED DESCRIPTION:
The aims of this study are to evaluate the safety and tolerability of single intravenous (IV) doses of GW856553 in healthy adult subjects and to investigate the relationship between PK and PD markers within the first few hours following administration of study drug to support progression of this formulation into a patient population.

Subjects in Cohort 1 (n=4) will receive a single 1mg IV dose (given as a 15 minute infusion) of GW856553. Safety, tolerability and PK exposures will be reviewed, and in an optional cohort (Cohort 2) (n=4), the dose may be adjusted upward or downward based on data from Cohort 1. Based on the results from Cohort 1 (and Cohort 2 if required), Cohort 3 (n=12) will be dosed appropriately to receive a single IV 15 minute infusion of GW856553.

After a one week washout, Cohort 3 subjects will receive a single oral dose of 15mg GW856553. Access to both IV and oral PK in the same individuals will permit calculation of absolute bioavailability for the oral dose. Subjects will be resident in the research unit from the morning prior to dosing until after the last PK blood sample is collected at 24 hours after the dose of study drug (excluding any washout period).

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhoea
* Male subjects must agree to use contraception from the time of the first dose of study medication until seven days following the last dose.
* Body weight >50kg (110 pounds) and body mass index (BMI) within the range >19 and <30kg/m2.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125ml) of wine or 1 (25ml) measure of spirits.
* Treatment with an investigational product within 90 days or 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to dosing in this study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02-02 (Actual); Primary Completion 2010-04-15 (Actual); Study Completion 2010-04-15 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability endpoints include changes in clinical laboratory assessments, spontaneous AE reporting, ECGs, vital signs and nursing/physician observations. | Up to 15 days post IV infusion.

SECONDARY OUTCOMES:
pHSP27 measurements | Up to 24 hours post dose.
hsCRP measurements | Up to 24 hours post dose.
Maximum Plasma Concentration [Cmax] | Up to 24 hours post dose
Area Under the Curve [AUC] | Up to 24 hours post dose
Time of maximum plasma concentation [Tmax] | Up to 24 hours post dose
Half life [T1/2] | Up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Barbour AM, Sarov-Blat L, Cai G, Fossler MJ, Sprecher DL, Graggaber J, McGeoch AT, Maison J, Cheriyan J. Safety, tolerability, pharmacokinetics and pharmacodynamics of losmapimod following a single intravenous or oral dose in healthy volunteers. Br J Clin Pharmacol. 2013 Jul;76(1):99-106. doi: 10.1111/bcp.12063. PMID 23215699
- See also: Results for study 113022 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113022?search=study&search_terms=113022#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 113022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register